CLINICAL TRIAL: NCT01088113
Title: The Relationship Between Cranial Near-InfraRed Oxygenation(NIRO) and Heart Rate Variability During Mental Exercise
Status: Completed | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Prof. Alice Jones, The Hong Kong Polytechnic University
Other Study IDs: HSEARS20080828002
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2008-08

CONDITIONS: Tai Chi Practitioner; Qigong Practitioner
Keywords: Tai Chi; Qigong; Heart rate variability; Near Infrared Spectroscopy; blood pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Tai Chi: Healthy subjects with Tai Chi practice
- Qigong: Healthy subjects with Qigong practice

SUMMARY:
The objective of this study is to investigate the effect of Tai Chi and Qigong practice on cranial oxyhaemoglobin level, blood pressures and autonomic nervous system responses.

ELIGIBILITY:
Inclusion Criteria:

* A minimal of 3 years experience on practice of either Tai Chi or Qigong

Exclusion Criteria:

* Unable to communicate or follow an exercise protocol
* Presence of cognitive impairments
* Symptomatic cardiovascular diseases
* Hypertension
* Diagnosis of stroke
* Parkinson's disease, or other neurologic disorder, peripheral neuropathy and cancer.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Level of Oxyhaemoglobin and total Haemoglobin

SECONDARY OUTCOMES:
Heart rate variability

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiopulmonary and Exercise Physiology Laboratory, The Hong Kong Polytechnic University, Hong Kong, Hong Kong, China